CLINICAL TRIAL: NCT06134583
Title: Effect of Superior Cervical Sympathetic Block Versus Stellate Ganglion Block to Treat Cerebral Vasospasm in Patients With Refractory Post-traumatic Subarachnoid Hemorrhage.
Brief Title: Superior Cervical Sympathetic Block Versus Stellate Ganglion Block in Post-traumatic Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rabab Ahmed Samy Anwer, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSB in SAH
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Post-Traumatic Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage, Traumatic

STUDY DESIGN:
Intervention Model Description: Comparison between superior cervical sympathetic block and stellate ganglion block to treat cerebral vasospasm in post-traumatic subarachnoid hemorrhage
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trible masking (participant, care provider and outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superior cervical ganglion block group (CSB) (Active Comparator): standardized protocol + CSB
  Interventions: Procedure: Superior cervical sympathetic block group
- Stellate ganglion block group (SGB) (Active Comparator): standardized protocol + SGB
  Interventions: Procedure: Stellate ganglion block group

INTERVENTIONS:
Procedure: Superior cervical sympathetic block group — 5 ml bupivacaine 0.5% will be injected around the internal carotid artery at the level of carotid bifurcation
  Other Names: CSB
  Arms: Superior cervical ganglion block group (CSB)
Procedure: Stellate ganglion block group — 5 ml bupivacaine 0.5% will be injected between the common carotid artery and longus capitis muscle at the level of C7 vertebra
  Other Names: SGB
  Arms: Stellate ganglion block group (SGB)

SUMMARY:
Posttraumatic Subarachnoid hemorrhage (SAH) is a life-threatening neurological problem with a high mortality rate. Delayed cerebral ischemia (DCI) is the second-leading cause of death and disability in patients suffering from SAH. DCI is strongly associated with cerebral arterial vasospasm (CAV), which reduces cerebral blood flow (CBF) and causes cerebral infarction.

Various treatment modalities have been tried for the prevention and treatment of vasospasm, including oral nimodipine and isovolumic hypertension, as well as endovascular treatments such as intra-arterial drug infusion and balloon angioplasty. A few studies have demonstrated the role of stellate ganglion block (SGB) in the management of this dreaded complication.

Cervical sympathetic block (CSB) may be an effective therapy but is not routinely performed to treat vasospasm/DCI. CSB is a local, minimally invasive, low cost and safe technique that can be performed at the bedside and may offer significant advantages as complementary treatment in combination with more conventional neurointerventional surgery interventions.

Aim of study is evaluating the effect of superior sympathetic ganglion block versus stellate ganglion block in treating cerebral vasospasm and prevention of delayed cerebral ischemia in refractory post-traumatic subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Trauma patients with CT evidence of post-traumatic SAH will be enrolled in the study and randomly assigned into two groups (30 patients each):

1. Group A: Superior cervical ganglion block group (CSB); 5 ml bupivacaine 0.5% will be injected around the internal carotid artery at the level of carotid bifurcation on the side of spasm and on each side if bilateral spasm using USG.
2. Group B: Stellate ganglion block group (SGB); 5 ml bupivacaine 0.5% will be injected between the common carotid artery and longus capitis muscle at the level of C7 vertebra on the side of spasm and on each side if bilateral spasm using USG.

All patients will be treated with a standardized protocol that included immediate intensive care monitoring, hypertension (MABP < 90 mmHg) and avoidance of hypotensive events, fluid resuscitation to maintain hypervolemia (defined as a positive fluid balance >500 mL/d), and spontaneous hemodilution at 0.3 hematocrit. All patients will receive oral nimodipine for 3 weeks. Analgesia as needed and sedation will be avoided if possible.

Intervention Technique:

1. Superior cervical ganglion block technique;

   * Patients will be placed in the supine position with the head turned to the opposite side of injection.
   * Procedure will be done under complete aseptic technique; mastoid process, hairline, and neck will be disinfected.
   * The common carotid artery will be identified by a high resolution linear ultrasound probe.
   * The probe gradually moved in the cranial direction to the position of the carotid bifurcation.
   * The C2- vertebral transverse process, vertebral artery, longus capitis muscle (LCM), and sternocleidomastoid muscle have been located to determine the puncture route,
   * After injection of a local anesthetic to the skin a needle (25-G injection needle) will be introduced using the in-plane approach, and 5 mL solution of bupivacaine 0.5% will be injected just behind the internal carotid artery.
   * Monitoring during procedure, vital signs (blood pressure, ECG and SPO2) every 10 minutes up to 30 min after block.
   * Endpoints for procedure success are signs of Horner's syndrome will be examined up to 30 min after block.
   * Patients with failed SGB will be excluded.
2. Stellate ganglion block technique;

   * Patients will be placed in the supine position with the head turned to the opposite side of injection.
   * Procedure will be done under complete aseptic technique; mastoid process, hairline, and neck will be disinfected.
   * The posterior tubercle of C7 vertebrae, vertebral artery will be identified by a high resolution linear ultrasound probe.
   * The probe is moved medially opposite to the level of C7 identifying the common carotid artery, 5 ml solution of bupivacaine 0.5% will be injected between the common carotid and longus colli muscle.
   * The endpoint criterion of SGB success is Horner's syndrome, which is characterized by miosis, ptosis, enophthalmos, conjunctival hyperemia, and facial redness without sweating. The patient will be monitored for at least 30 min to rule out any related complications after SGB.
   * Patients with failed SGB will be excluded.
3. Basic Transcranial Doppler Exam; A low-frequency ultrasound probe is required (2-3 MHz) due to improved penetration of ultrasound waves through the cranial temporal bones. Both the power M-mode and Doppler mode will be utilized transtemporal window will be used to assess circle of wills arteries.

Transtemporal window:

1. MCA: Depth of 45-65mm with direction toward the probe.
2. MCA/ACA bifurcation: Depth of 60-65mm with bidirectional flow.
3. ACA: Depth of 60-75mm with direction away from the probe.
4. PCA (P1): Depth of 60-75mm with direction toward the probe.
5. PCA (P2): Depth of 60-75mm with direction away from the probe.
6. Terminal ICA: Depth of 60-65mm with direction toward the probe.

Parameters extracted from TCD:

1. Mean cerebral blood flow velocity: Calculated using peak systolic velocity (PSV) and end-diastolic velocity (EDV) based on the following formula: [PSV + (EDV x 2)]/3[1].
2. Resistive index: Measure of resistance to blood flow. RI = (PSV - EDV)/PSV[8].
3. Lindegaard ratio (LR): The LR is a calculated value that normalizes the MCA velocity to the ICA. This is calculated by the mean velocity of the MCA divided by the mean velocity of the ICA. This ratio is important for differentiating hyperemia from true vasospasm on TCD study. If the MCA is increased at a higher proportion than the ICA, it indicates vasospasm as the source of the elevated velocity. A normal LR is considered < 3, mild vasospasm 3.0-4.5, moderate vasospasm 4.5-6.0 and severe vasospasm >6.0.

Pre-interventional Parameters evaluation: -

Standard monitoring includes:

* Hemodynamics [ECG, Spo2, SBP, DBP and MBP] every 10 minutes during procedure upto 30 minutes after block.
* Arterial oxygen saturation.
* Continuous invasive arterial blood pressure monitoring (IABP): systolic arterial blood pressures (SABP), diastolic arterial blood pressure (DABP), mean arterial blood pressure (MABP).
* Temperature.
* Preintervention assessment of GCS, CBF by TCD assessment of MCA, ACA and LR ratio and cerebral blood vessels diameter by MRA whenever possible.

Post-interventional data collection: -

* Duration of study: 24 hours after intervention.
* Hemodynamics; HR and MBP every 10 minutes up to 2h after block and then every hour.
* Postintervention reassessment of CBF by TCD assessment of MCA, ACA and LR ratio by the same observer 30 minutes, 6 hours, 24 hours after block.
* Cerebral blood vessels diameter by MRA within the first 4 hours after block whenever possible.
* Any change in GCS within 24h after block.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patient with radiological evidence of refractory SAH despite adequate pharmacological treatment; TCD velocity > 120 cm/sec.
* Trauma Patients with clinicoradiological evidence of cerebral vasospasm. The clinical criteria is new onset of neurological impairment such as hemiparesis, aphasia, hemianopia, or decrease of at least 2 points on the GCS not explained by appearance of new finding in follow up CT.
* Age 18-65 will be included in the study
* Both sex are included .

Exclusion Criteria:

* Refusal to consent participating research from patient or his guardian.
* Patients with deterioration in the level of consciousness due to other causes such as rebleeding, infarct, hydrocephalus, cerebral edema, infection, electrolyte disorder, or seizure.
* Trauma and local infection in the nerve block area.
* Coagulopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
TCD velocities | 24 hours
  changes in transcranial Doppler (TCD) velocities of middle cerebral artery (MCA) before and after block.

SECONDARY OUTCOMES:
New vasospasm | 24 hours
  The incidence of new TCD vasospasm and new CT cerebral infarction.
GCS | 24 hours
  Changes in Glasgow Coma Scale (GCS) after block.
Technical complications | 24 hours
  Incidence of technical complications.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Campos-Pires R, Edge CJ, Dickinson R. Argon: A Noble Foe for Subarachnoid Hemorrhage. Crit Care Med. 2016 Jul;44(7):1456-7. doi: 10.1097/CCM.0000000000001680. No abstract available. PMID 27309177
- [Result] Dodd WS, Laurent D, Dumont AS, Hasan DM, Jabbour PM, Starke RM, Hosaka K, Polifka AJ, Hoh BL, Chalouhi N. Pathophysiology of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage: A Review. J Am Heart Assoc. 2021 Aug 3;10(15):e021845. doi: 10.1161/JAHA.121.021845. Epub 2021 Jul 30. PMID 34325514
- [Result] Abboud T, Andresen H, Koeppen J, Czorlich P, Duehrsen L, Stenzig J, Westphal M, Regelsberger J. Serum levels of nimodipine in enteral and parenteral administration in patients with aneurysmal subarachnoid hemorrhage. Acta Neurochir (Wien). 2015 May;157(5):763-7. doi: 10.1007/s00701-015-2369-9. Epub 2015 Feb 21. PMID 25701099
- [Result] Kosnik EJ, Hunt WE. Postoperative hypertension in the management of patients with intracranial arterial aneurysms. J Neurosurg. 1976 Aug;45(2):148-54. doi: 10.3171/jns.1976.45.2.0148. PMID 939973
- [Result] Raabe A, Beck J, Keller M, Vatter H, Zimmermann M, Seifert V. Relative importance of hypertension compared with hypervolemia for increasing cerebral oxygenation in patients with cerebral vasospasm after subarachnoid hemorrhage. J Neurosurg. 2005 Dec;103(6):974-81. doi: 10.3171/jns.2005.103.6.0974. PMID 16381183
- [Result] Cho WS, Kang HS, Kim JE, Kwon OK, Oh CW, Son YJ, Know BJ, Jung C, Hang MH. Intra-arterial nimodipine infusion for cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage. Interv Neuroradiol. 2011 Jun;17(2):169-78. doi: 10.1177/159101991101700205. Epub 2011 Jun 20. PMID 21696654
- [Result] Jain V, Rath GP, Dash HH, Bithal PK, Chouhan RS, Suri A. Stellate ganglion block for treatment of cerebral vasospasm in patients with aneurysmal subarachnoid hemorrhage - A preliminary study. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):516-21. doi: 10.4103/0970-9185.86598. PMID 22096287
- [Result] Bombardieri AM, Albers GW, Rodriguez S, Pileggi M, Steinberg GK, Heit JJ. Percutaneous cervical sympathetic block to treat cerebral vasospasm and delayed cerebral ischemia: a review of the evidence. J Neurointerv Surg. 2023 Dec;15(12):1212-1217. doi: 10.1136/jnis-2022-019838. Epub 2022 Dec 6. PMID 36597947
- [Result] Maeda A, Chikama Y, Tanaka R, Tominaga M, Shirozu K, Yamaura K. Safety and utility of ultrasound-guided superior cervical ganglion block for headaches and orofacial pain: a retrospective, single-center study of 10 patients. JA Clin Rep. 2023 Apr 29;9(1):21. doi: 10.1186/s40981-023-00613-z. PMID 37119368
- [Result] Jing L, Wu Y, Liang F, Jian M, Bai Y, Wang Y, Liu H, Wang A, Chen X, Han R. Effect of early stellate ganglion block in cerebral vasospasm after aneurysmal subarachnoid hemorrhage (BLOCK-CVS): study protocol for a randomized controlled trial. Trials. 2022 Nov 4;23(1):922. doi: 10.1186/s13063-022-06867-9. PMID 36333751